CLINICAL TRIAL: NCT04234217
Title: Mechanisms of Prediabetic States in Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Mayo Clinic (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB19-0593; R01HL146127 (NIH)
Record Dates: First submitted 2019-12-18; First posted 2020-01-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea; Pre-diabetes
Keywords: Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Glucose Intolerance | interventions — Continuous Positive Airway Pressure; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Untreated (No Intervention): Untreated condition (obstructive sleep apnea)
- Continuous positive airway pressure (CPAP) treatment (Active Comparator): Continuous positive airway pressure (CPAP) treatment
  Interventions: Device: Continuous positive airway pressure
- Niacin (Active Comparator): Untreated, pharmacological suppression of lipolysis by Niacin
  Interventions: Other: Niacin

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure (CPAP) treatment of obstructive sleep apnea (OSA)
  Other Names: CPAP
  Arms: Continuous positive airway pressure (CPAP) treatment
Other: Niacin — Suppression of lipolysis by niacin infusion
  Other Names: Suppression of lipolysis by niacin infusion
  Arms: Niacin

SUMMARY:
The purpose of this study is to better understand how sleep apnea contributes to the development of diabetes.

DETAILED DESCRIPTION:
Substantial evidence indicates that obstructive sleep apnea (OSA) is associated with impaired glucose metabolism, however, metabolic mechanisms underlying this association remain unclear. This mechanistic study will determine systemic and cellular metabolic pathways that contribute to impaired glucose metabolism in obstructive sleep apnea (OSA). Understanding of how obstructive sleep apnea (OSA) affects glucose metabolism may help identify novel targets for risk prediction and/or treatment of metabolic impairments beyond continuous positive airway pressure (CPAP). Obstructive sleep apnea (OSA) patients with prediabetes will be studied under three in-laboratory conditions in a randomized cross-over design: untreated condition (obstructive sleep apnea), treated condition (continuous positive airway pressure), untreated but pharmacologically suppressed lipolysis condition (Niacin). The investigator will perform whole body and cellular assessments under each study condition.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Prediabetic
* Sleep apnea

Exclusion Criteria:

* Diabetic
* Severe hypertension
* Taking medications that can confound assessments
* Any history of known bleeding disorders
* Any underlying disease likely to limit life span or increase risk of intervention
* Currently pregnant, trying to get pregnant or nursing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Plasma norepinephrine levels | Untreated, within 4 months of screening
  Plasma norepinephrine will be measured in blood
Plasma norepinephrine levels | CPAP, within 4 months of screening
  Plasma norepinephrine will be measured in blood
Plasma norepinephrine levels | Niacin, within 4 months of screening
  Plasma norepinephrine will be measured in blood

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No